CLINICAL TRIAL: NCT00976729
Title: NOX-E36 - A Phase I, Double-Blind, Placebo Controlled, Single Intravenous and Subcutaneous Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Healthy Subjects
Brief Title: NOX-E36 First-in-Human (FIH) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNOXE36C001
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Inflammatory Diseases; Type 2 Diabetes Mellitus; Systemic Lupus Erythematosus
Keywords: monocyte chemoattractant protein-1 (MCP-1); L-oligonucleotide aptamer; Spiegelmer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Placebo i.v. (Placebo Comparator)
  Interventions: Drug: Placebo
- 0.03 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- 0.09 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- 0.25 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- 0.5 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- 1.0 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- 2.0 mg/kg i.v. (Experimental)
  Interventions: Drug: NOX-E36
- Placebo s.c. (Placebo Comparator)
  Interventions: Drug: Placebo
- 0.25 mg/kg s.c. (Experimental)
  Interventions: Drug: NOX-E36
- 0.5 mg/kg s.c. (Experimental)
  Interventions: Drug: NOX-E36

INTERVENTIONS:
Drug: NOX-E36 — single ascending IV doses, ranging from 0.03 mg/kg to 2.0 mg/kg
  Arms: 0.03 mg/kg i.v.; 0.09 mg/kg i.v.; 0.25 mg/kg i.v.; 0.5 mg/kg i.v.; 1.0 mg/kg i.v.; 2.0 mg/kg i.v.
Drug: NOX-E36 — single SC doses, at safe and tolerable dose level
  Arms: 0.25 mg/kg s.c.; 0.5 mg/kg s.c.
Drug: Placebo
  Arms: Placebo i.v.; Placebo s.c.

SUMMARY:
This is the first time NOX-E36 will be administered to man. The principal aim of this study is to obtain safety and tolerability data when NOX-E36 is administered by single intravenous (IV) and subcutaneous (SC) doses to healthy male and female subjects. This information, together with the pharmacokinetic and pharmacodynamic data, will help establish the doses, dosage regimen and route of administration suitable for multiple dose administration to healthy volunteers, followed by the studies in the patient population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Body mass index (BMI) between 19.0 and 29.0 kg/m2 inclusive
* Body weight between 50 and 100 kg inclusive
* Creatinine clearance of greater than 80 mL/min

Exclusion Criteria:

* Male and female subjects who are not or whose partners are not willing to use appropriate contraception methods
* Intake of any prescribed systemic or topical medication within 14 days prior to dosing
* Intake of any non-prescribed systemic or topical medication (including herbal remedies) within 7 days prior to dosing (with the exception of vitamin/mineral supplements)
* Supine blood pressure and supine pulse rate higher than 140/90 mmHg and 100 beats per minute (bpm), respectively, or lower than 90/50 mmHg and 40 bpm, respectively, as confirmed by a repeat assessment
* History of any clinically significant neurological, dermatological, gastrointestinal, renal, hepatic, cardiovascular, psychiatric, respiratory, metabolic, endocrine, haematological or other major disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NOX-E36 by means of adverse events, vital signs, laboratory parameters, 12-lead ECG and immunogenicity assessment | throughout the entire study

SECONDARY OUTCOMES:
Pharmacokinetic parameters in plasma and urine | throughout the entire study
Pharmacodynamic profile | throughout the entire study

CONTACTS AND LOCATIONS:
Overall Officials: Grit Landgraf, PhD, Study Director — Noxxon AG